CLINICAL TRIAL: NCT06395194
Title: The Valsartan Antihypertensive Long-term Use Evaluation Trial
Brief Title: Effects of Valsartan vs Amlodipine and Low BP on Kidney Outcomes in Essential Hypertension
Acronym: VALUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Sverre Erik Kjeldsen, Professor Emeritus, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OsloUHtheValueTrial
Record Dates: First submitted 2024-04-10; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Essential Hypertension
Keywords: Hypertension; Blood pressure; valsartan; amlodipine; kidney disease
MeSH Terms: conditions — Essential Hypertension; Hypertension; Kidney Diseases | interventions — Valsartan; Angiotensin Receptor Antagonists; Amlodipine; Calcium Channel Blockers

STUDY DESIGN:
Intervention Model Description: Investigator-designed, prospective, multi-national, double-blind, randomized, active-controlled, parallel-group design which was event driven (until accumulated 1450 primary cardiac endpoints)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Preparation of the two drugs (to compare, valsartan and amlodipine) made identical
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Valsartan (Active Comparator): Treatment based on the ARB valsartan
  Interventions: Drug: Cardiac outcomes on treatment with valsartan
- Amlodipine (Active Comparator): Treatment based on the CCB amlodipine
  Interventions: Drug: Cardiac outcomes on treatment with amlodipine

INTERVENTIONS:
Drug: Cardiac outcomes on treatment with valsartan — Patients who already were on treatment, discontinued their previous antihypertensive medications when randomized to one of the trial's masked study arms (valsartan or amlodipine) without a run-in phase ("rolled over"). Valsartan treatment started at a dosage of 80 mg daily. If BP did not reach <140/90 mmHg, the valsartan dose was doubled to 160 mg, and then hydrochlorothiazide (12.5 mg and 25 mg daily) and other antihypertensive drugs were added in sequential steps.
  Other Names: Angiotensin-receptor blocker
  Arms: Valsartan
Drug: Cardiac outcomes on treatment with amlodipine — Patients who already were on treatment, discontinued their previous antihypertensive medications when randomized to one of the trial's masked study arms (valsartan or amlodipine) without a run-in phase ("rolled over"). Amlodipine treatment started at 5 mg daily. If BP did not reach <140/90 mmHg, the amlodipine dose was doubled to 10 mg, and then hydrochlorothiazide (12.5 mg and 25 mg daily) and other antihypertensive drugs were added in sequential steps.
  Other Names: Calcium-channel blocker
  Arms: Amlodipine

SUMMARY:
The Valsartan Antihypertensive Long-term Use Evaluation (VALUE) trial tested the hypothesis that for the same blood-pressure control, valsartan would reduce cardiac morbidity and mortality more than amlodipine in hypertensive patients at high cardiovascular risk. The present study investigates effects of valsartan and amlodipine on pre-specified secondary kidney outcomes.

DETAILED DESCRIPTION:
VALUE was a multicenter, prospective, double-blinded randomized clinical trial initiated and led by the investigators. The study took place from 1997 to 2004. The sponsor was Novartis, who had an interactive role with the investigators for the study design, and Novartis monitored study sites and provided source data verifications. In 2011, Ullevaal University Hospital, Oslo, Norway, took over the database with conditions detailed in a written agreement with the funder. One author (S.E.K.) had from then full access to all the data and took responsibility for its integrity and the data analysis. Thus, the data file resides in the hands of the authors, and Novartis had no role in the present study.

The trial was approved by ethics committees and written informed consent collected from all the participants in 31 countries.

The study compared, in a prospective, randomized double-blinded design, the effects of two different antihypertensive treatment regimens on cardiac morbidity and mortality in hypertensive patients aged 50 years or older. One regimen was based on the ARB valsartan, and the other on the CCB amlodipine.

VALUE participants were selected based on predefined combinations of risk factors, including age, male gender, and the presence of certain conditions such as electrocardiographic left ventricular hypertrophy (ECG-LVH), determined by Cornell voltage-duration product or Sokolow-Lyon voltage criteria with or without a strain pattern, serum creatinine ≥150 μmol/l, proteinuria (positive dipstick in morning urine at two different visits), diabetes mellitus (DM), or verified coronary, cerebrovascular, or peripheral artery disease.

Exclusion criteria included pregnancy, renal artery stenosis, either myocardial infarction, percutaneous coronary intervention, or coronary artery bypass surgery during last three months, medically relevant valvular disease, cerebrovascular events last 3 months, severe hepatic disease, severe chronic kidney failure (serum creatinine >3.0 mg/dl, >265 µmol/L), congestive heart failure requiring angiotensin converting enzyme inhibitor and patients using beta-blocker for both coronary artery disease and hypertension.

Participants were followed for 4-6 years, until a minimum of 1450 primary cardiac events ("endpoint driven") with monthly visits during the initial six months after randomization and later at six-month intervals. BP was measured at each visit using a calibrated sphygmomanometer or a validated digital device with an appropriate size cuff. Patients were seated quietly for 5 minutes before the measurement of BP. Blood samples were collected and analyzed at central labs in each continent. Serum creatinine was measured yearly.

The primary goal of the study was to determine the time to the occurrence of the first cardiac event, which included a combination of fatal or non-fatal myocardial infarction, sudden cardiac death, death from revascularization procedures or heart failure, hospitalization for heart failure, and emergency procedures to prevent myocardial infarction. The secondary endpoints were all cardiovascular events, fatal and non-fatal stroke, myocardial infarction, hospitalized heart failure, cardiovascular-, non-cardiovascular-, and all-cause mortality.

Pre-specified secondary kidney endpoints were end-stage kidney disease (ESKD) in patients with need for dialysis or kidney transplantation and worsened kidney function (WKF) with at least 50% increase in serum creatinine from baseline. To ensure impartiality, the endpoint committee was not informed of the treatment assignments when assessing events.

Patients who were previously treated for hypertension (92%) were eligible if SBP was <210 mmHg and diastolic(D) BP was <115 mmHg. Untreated hypertensive patients were eligible if SBP was between 160 and 210 mmHg, and DBP was <115 mmHg. Patients who already were on treatment, discontinued their previous antihypertensive medications when randomized to one of the trial's masked study arms (valsartan or amlodipine) without a run-in phase ("rolled over"). Valsartan treatment started at a dosage of 80 mg daily, and amlodipine treatment started at 5 mg daily. If BP did not reach <140/90 mmHg, the dose of either drug was doubled to 160 mg or 10 mg, respectively, and hydrochlorothiazide (12.5 mg and 25 mg daily) and other antihypertensive drugs were added in sequential steps.

Age, the presence of coronary heart disease, and the presence of ECG-LVH at baseline were used in the randomized study as à priori covariates to account for the effects of key risk predictors at baseline.

To minimize the influence of potential confounding factors, hazard ratios (HRs) in the observational analysis of different achieved BP levels were adjusted for treatment allocation and baseline covariates including age, sex, SBP, diastolic blood pressure, body mass index, smoking status, high serum total cholesterol (>6.2 mmol/L or >240 mg/dL), presence of diabetes mellitus, proteinuria, ECG-LVH, previous stroke, previous myocardial infarction, and previous peripheral artery disease.

Statistical power was calculated for the original comparison of valsartan vs amlodipine on the primary endpoint.15 The trial was endpoint driven, needed 1450 primary events to close, and showed no difference between valsartan and amlodipine on the primary endpoint, which allowed consolidation of data from both treatment arms for other studies of this hypertensive population like investigation BP variability and the influence of achieved BPs on certain endpoints. Of the 15,245 hypertensive patients enrolled by 969 investigators, 13,803 patients did not experience any cardiovascular event during the initial six months of treatment after randomization and had attended a minimum of three study visits after that period. A minimum of three visits was decided à priori to ensure meaningful follow up of representative achieved BPs. Patients with cardiovascular events during the first six months after randomization were excluded because of the uncontrolled BP following discontinuation of previous antihypertensive drugs and concomitant up-titration of the randomized medications; these early BPs were neither included as they were not representative for the later achieved average BPs.

Treatment effects on kidney endpoints in the RCT were measured by hazard ratios and their 95% CIs based on Cox regression models and analyzed as intention-to-treat. Event rates over time are presented as Kaplan-Meier curves. Similar multivariate adjusted Cox models were used to analyze the kidney endpoints for patients who achieved average SBP <135 mmHg vs SBP ≥135 mmHg up to the occurrence of a prespecified endpoint, or throughout the treatment period if no event occurred. Similar comparisons were done for patients who achieved average DBP <85 mmHg vs ≥85 mmHg and for groups with SBP ≥135 and/or DBP ≥85 mmHg vs patients with SBP <135 and DBP <85 mmHg.

Statistical significance was determined with a two-sided p-value of <0.05. Data analysis was carried out using SPSS (IBM SPSS Statistics: Version: 28.0.1.0, Armonk, NY, USA). Data are presented as means with standard deviations (SDs), absolute numbers with percentages in parentheses, or point estimates with 95% confidence intervals (CIs).

ELIGIBILITY:
Inclusion Criteria:

* hypertension, and predefined combinations of risk factors, including:
* age
* male gender
* the presence of electrocardiographic left ventricular hypertrophy (LVH, determined by Cornell voltage-duration product or Sokolow-Lyon voltage criteria with or without a strain pattern)
* serum creatinine ≥150 μmol/l
* proteinuria (positive urine dipstick at two occasions)
* type 2 diabetes mellitus
* verified coronary, cerebrovascular, or peripheral artery disease

Exclusion Criteria:

* pregnancy
* renal artery stenosis
* myocardial infarction, percutaneous coronary intervention, or coronary artery bypass surgery during last three months
* medically relevant cardiac valvular disease
* cerebrovascular events last 3 months
* severe hepatic disease
* severe chronic kidney failure (serum creatinine >3.0 mg/dl, >265 µmol/L)
* congestive heart failure requiring angiotensin converting enzyme inhibitor (ACEI)
* use of beta-blocker for both coronary artery disease and hypertension

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15313 (Actual)
Dates: Start 1997-09-27 (Actual); Primary Completion 2003-09-05 (Actual); Study Completion 2003-12-05 (Actual)

PRIMARY OUTCOMES:
Composite cardiac event (mostly myocardial infarction and heart failure hospitalization) | Up to 6 years
  Composite cardiac events, which included a combination of fatal or non-fatal myocardial infarction, sudden cardiac death, death from revascularization procedures or heart failure, hospitalization for heart failure, and emergency procedures to prevent myocardial infarction

SECONDARY OUTCOMES:
End-stage kidney failure | Up to 6 years
  Incident end-stage kidney disease being patients in need for dialysis or kidney transplantation
Worsened kidney function | Up to 6 years
  No of patients with at least 50% increase of serum creatinine.
All cardiovascular events | Up to 6 years
  All cardiovascular events
Stroke | Up to 6 years
  Fatal and non-fatal stroke
Myocardial infarction | Up to 6 years
  Fatal and non-fatal myocardial infarction
Heart failure | Up to 6 years
  Hospitalized for heart failure
Cardiovascular mortality | Up to 6 years
  All deaths from cardiovascular disease
Non-cardiovascular mortality | Up to 6 years
  All deaths from causes other than cardiovascular disease
All-cause mortality | Up to 6 years
  All deaths during folllow-up, from all causes

CONTACTS AND LOCATIONS:
Overall Officials: Sverre E Kjeldsen, MD, PhD, Study Chair — University Of Oslo Hospital

IPD SHARING:
Plan to Share IPD: No
Partial IPD sharing with the BPLTTC Group in Oxford

REFERENCES:
- [Result] Julius S, Kjeldsen SE, Weber M, Brunner HR, Ekman S, Hansson L, Hua T, Laragh J, McInnes GT, Mitchell L, Plat F, Schork A, Smith B, Zanchetti A; VALUE trial group. Outcomes in hypertensive patients at high cardiovascular risk treated with regimens based on valsartan or amlodipine: the VALUE randomised trial. Lancet. 2004 Jun 19;363(9426):2022-31. doi: 10.1016/S0140-6736(04)16451-9. PMID 15207952
- [Derived] Olsen E, Soraas CL, Schmieder RE, Jamerson K, MacDonald TM, Mancia G, Heimark S, Mehlum MH, Liestol K, Larstorp ACK, Mariampillai JE, Mo R, Halvorsen LV, Hoieggen A, Rostrup M, Kjeldsen SE, Weber MA. Low Achieved Systolic Blood Pressure Related to Kidney Protection in Diabetic and Non-Diabetic High-Risk Hypertensive Patients. Am J Hypertens. 2025 Nov 17;38(12):1106-1119. doi: 10.1093/ajh/hpaf093. PMID 40397037